CLINICAL TRIAL: NCT00711633
Title: Evaluation of a Fermented Formula Without Live Bacteria for Preterm Infants: Effects on Microbiota Species and Intestinal Inflammatory Markers
Brief Title: Evaluation of Safety, Tolerance and Effects on the Intestinal Flora of a New Fermented Milk for Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Blédina SA, Villefranche sur Saône, France (Unknown)
Responsible Party: Serreau, URC Paris Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1977/06-05-02
Record Dates: First submitted 2008-07-04; First posted 2008-07-09 (Estimated); Last update posted 2008-07-09 (Estimated); Status verified 2008-06

CONDITIONS: Preterms With Gestational Age Ranging From 30 to 35 Weeks
Keywords: Premature birth,; infant,; infant formula,; bacterial colonization,; Bifidobacterium,; calprotectin
MeSH Terms: conditions — Premature Birth | interventions — Milk; Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): the fermented preterm formula (FPF)
  Interventions: Dietary Supplement: Milk with probiotic and prebiotic activities
- 2 (Placebo Comparator): formula adapted for preterm infants (PF)
  Interventions: Dietary Supplement: Milk without probiotic and prebiotic activities

INTERVENTIONS:
Dietary Supplement: Milk with probiotic and prebiotic activities — Comparison of two different formula for preterm infants
  Arms: 1
Dietary Supplement: Milk without probiotic and prebiotic activities — Comparison of formula for preterm infants
  Other Names: Comparison of formula for preterm infants
  Arms: 2

SUMMARY:
The intestinal flora is a complex ecosystem which is known to play various important functions in the gut. Recent data have reported a delay in intestinal colonization in preterm. Modulating the intestinal flora through dietary supplementation with probiotics or prebiotics has been shown to improve digestive and general outcomes in full-term infants.The aim of this study was to evaluate the clinical tolerance, the effect on gut microbiota, and the mucosal inflammatory responses to a fermented milk in preterm infants.

DETAILED DESCRIPTION:
This prospective, randomized, double-blind, controlled study evaluated the safety and effect on gut microbiota, and the mucosal inflammatory responses to a fermented milk in preterm infants. Preterm infants with a gestational age (GA) ranging from 30 to 35 weeks and whose mother chose formula feeding were enrolled during their first three days of life. Both parents provided informed written consent. Infants were randomly assigned to receive either the fermented preterm formula (FPF) or, as a control, a formula adapted for preterm infants (PF). The PF was formulated to meet the nutritional needs of preterm infants. The FPF was identical, except for a manufacturing process including a fermentation step with two probiotic strains, Bifidobacterium breve C50 and Streptococcus thermophilus 065, inactivated by heat at the end of the manufacturing process. This process conferred a probiotic/prebiotic activity.For each neonate, background information about the pregnancy and neonatal parameters were collected. Anthropometric parameters (weight, height, head circumference); gastrointestinal tolerance parameters (abdominal distension, gastric residuals, rectal bleeding, NEC); drug administration; and intake of formula and mother's milk were recorded twice a week until discharge. Stools were collected twice a week from diapers for microbiological analysis and measurement of fecal inflammatory markers. All samples were immediately stored at -80°C.

ELIGIBILITY:
Inclusion Criteria:

* Preterms with gestational age ranging from 30 to 35 weeks
* Eutrophic
* Formula feeding

Exclusion Criteria:

* Malformation or metabolic disease
* Newborns whose parents did not provide informed consent
* Contraindication to enteral feeding

Ages: 1 Day to 15 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2002-12; Primary Completion 2005-02 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Follow-up of the number of colonized infants and the bacterial colonization levels | weekly until hospital discharge

SECONDARY OUTCOMES:
Clinical tolerance | weekly until hospital discharge
Levels of intestinal immune and inflammatory markers | weekly until hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Florence Campeotto, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Neonatat unit, Saint Vincent de Paul Hospital, Paris, France

REFERENCES:
- [Background] Campeotto F, Waligora-Dupriet AJ, Doucet-Populaire F, Kalach N, Dupont C, Butel MJ. [Establishment of the intestinal microflora in neonates]. Gastroenterol Clin Biol. 2007 May;31(5):533-42. doi: 10.1016/s0399-8320(07)89424-3. French. PMID 17541346